CLINICAL TRIAL: NCT00013520
Title: Phase III, Randomized, Double-Blind Comparison of Three Protease Inhibitor-Sparing Regimens for the Initial Treatment of HIV Infection
Brief Title: Comparison of Three Different Initial Treatments Without Protease Inhibitors for HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5095; 10212 (Registry Identifier: DAIDS ES); ACTG A5095; AACTG A5095; Substudy ACTG A5097s; Substudy AACTG 5107s; Substudy AACTG 5166s; Substudy ACTG A5166s; Substudy AACTG 5097s; Substudy ACTG A5107s; 5K24AI051966-03 (NIH)
Record Dates: First submitted 2001-03-16; First posted 2001-08-31 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: HIV-1; Didanosine; Drug Therapy, Combination; Zidovudine; Nevirapine; Stavudine; Lamivudine; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Combivir; BMS 232632; Efavirenz; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine; Atazanavir Sulfate; lamivudine, zidovudine drug combination; efavirenz; Nevirapine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Abacavir sulfate, Lamivudine and Zidovudine
Drug: Atazanavir
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate
Drug: Efavirenz
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare the effectiveness, safety, and tolerability of 3 anti-HIV combination treatments that do not use protease inhibitors (PIs).

The current rule for starting treatment of HIV infection is to combine members from different classes of anti-HIV drugs, such as 2 nucleoside reverse transcriptase inhibitors (NRTIs) and either a PI or a nonnucleoside reverse transcriptase inhibitor (NNRTI). However, these combinations can be complicated and difficult to take, can cause a number of side effects, and may become ineffective. Combinations that are simpler, better tolerated, and more effective are needed. Because PIs can cause long-term side effects and because HIV can become resistant to many of them at the same time, anti-HIV combination treatments that do not use PIs are being tested.

DETAILED DESCRIPTION:
Current treatment guidelines recommend combination regimens of 2 nucleoside analogues with either a PI or an NNRTI for the initial treatment of HIV infection. However, the efficacy of current regimens is limited by their complexity, pharmacokinetic characteristics, short- and long-term side effects, and drug-resistance profiles at the time of virologic failure. Consequently, the identification of new initial regimens that are simpler, better tolerated, preserve treatment options in the event of failure, and improve antiretroviral potency is needed. In addition, recent concern over the long-term toxicities of PIs and the extensive cross-resistance among the available PIs have led to the testing of PI-sparing regimens.

Participants will be in this study for a minimum of 120 weeks and a maximum of approximately 4 years. In Step 1, patients are randomly selected to receive 1 of 3 blinded treatment regimens: abacavir (ABC)/lamivudine (3TC)/zidovudine (ZDV)/efavirenz (EFV), ABC/3TC/ZDV, or 3TC/ZDV/EFV. Patients with confirmed virologic failure on Step 1 and two successive plasma HIV RNA levels of 10,000 copies/ml or greater must register to Step 2. Patients with confirmed virologic failure on Step 1 and whose plasma HIV RNA is under 10,000 copies/ml may remain on Step 1 or register to Step 2. [AS PER AMENDMENT 04/11/03: Discontinuation of Arm B was recommended. Consequently, Arms A and C were unblinded to EFV but not to ABC. A number of options are available for patients originally randomized to Arm B.]

Step 2 is open label. Regimens include 2 or 3 nucleoside reverse transcriptase inhibitors (NRTIs) in combination with EFV, atazanavir (ATZ), ritonavir-boosted ATZ, or tenofovir disoproxil fumarate (TDF). Patients on Arm B treatment who have an HIV RNA level less than 200 copies/ml within the past 8 weeks are eligible for randomization to open-label intensification of Arm B on Step 3.

Step 3 regimens include ABC/3TC/ZDV plus either EFV or TDF. Patients with evidence of treatment-limiting toxicity to Step 3 study drugs have the option of substituting d4T for ZDV, ddI for ABC or TDF, and/or NVP for EFV. Patients with confirmed virologic failure on Step 3 and whose plasma HIV RNA is less than 10,000 copies/ml may either remain on Step 3 or register to Step 4. Patients with two successive plasma HIV RNA levels of 10,000 copies/ml or greater on Step 3 must register to Step 4.

Step 4 is open label. Regimens include two or three NRTIs plus EFV, ATV, ritonavir-boosted ATV, or TDF. Clinical assessments and laboratory evaluations are done at entry, at Weeks 2, 4, 6, 8, 12, 16, 20, 24, and then every 8 weeks thereafter for the duration of the study. Evaluations are also required when a protocol-allowed drug substitution is made.

In addition, 3 substudies are being conducted: a neurology substudy for efavirenz, a pharmacology substudy for atazanavir, and a viral dynamics substudy.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load of at least 400 copies/ml within 90 days prior to study entry.
* Are at least 16 years old.
* Weigh at least 40 kg.
* Have a negative pregnancy test within 48 hours before starting study drugs, if female and able to have children.
* Agree to use 2 effective methods of birth control while taking, and for 3 months after stopping, the study medications.
* Provide written consent of a parent or guardian, if under 18 years of age.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken anti-HIV drugs in the past.
* Are allergic to any of the study drugs or ingredients.
* Are pregnant or breast-feeding.
* Have taken any of the following drugs within 14 days prior to study entry: amiodarone, astemizole, bepridil, cisapride, ergot or ergot derivatives, systemic itraconazole, systemic ketoconazole, midazolam, propoxyphene, quinidine, rifampin, terfenadine, thalidomide, triazolam, or St. John's wort.
* Have taken drugs that influence the immune system, HIV or other vaccines, or investigational drugs within 30 days prior to study entry. Prednisone at a dose of 10 mg or less daily is allowed.
* Have taken drugs or been hospitalized for serious infections or medical illnesses within 14 days prior to study entry.
* Have growths or tumors that require drug therapy.
* Have Pneumocystis carinii pneumonia that is not clinically stable and whose treatment is not completed at least 7 days prior to study entry.
* Have infections or medical illnesses that are not under control or that have not received complete treatment before study entry.
* Have any condition that, in the opinion of the investigator, would prevent them from properly participating in the study.
* Abuse drugs or alcohol.
* This study has been updated to exclude patients who are receiving systemic itraconazole and rifabutin.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1125
Dates: Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Gulick, MD, Study Chair; Cecilia Shikuma, MD, Study Chair
Locations (60):
- United States (59):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Willow Clinic A0507 CRS, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - SSTAR, Family Healthcare Ctr., Fall River, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell CRS, New York, New York
  - Columbia Univ., HIV Prevention and Treatment Medical Ctr., New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - AIDS Care CRS, Rochester, New York
  - McCree McCuller Wellness Ctr. at the Connection, Infectious Disease Unit, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Philadelphia Veterans Admin. Med. Ctr. A6205 CRS, Philadelphia, Pennsylvania
  - Univ. of Pennsylvania Health System, Presbyterian Med. Ctr., Philadelphia, Pennsylvania
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Rhode Island Hosp., Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] H Ribaudo, D Clifford, R Gulick, C Shikuma, K Klingman, S Snyder, and E Acosta. Relationships between Efavirenz Pharmacokinetics, Side Effects, Drug Discontinuation, Virologic Response, and Race: Results from ACTG A5095/A5097s. CROI 2004. Abstract 132.
- [Result] Feinberg J. Meeting notes from the 2nd International AIDS Society Conference on HIV Pathogenesis and Treatment. Trizivir vs. efavirenz: results from ACTG 5095. AIDS Clin Care. 2003 Sep;15(9):78-9. PMID 14669723
- [Result] Gulick RM, Ribaudo HJ, Shikuma CM, Lustgarten S, Squires KE, Meyer WA 3rd, Acosta EP, Schackman BR, Pilcher CD, Murphy RL, Maher WE, Witt MD, Reichman RC, Snyder S, Klingman KL, Kuritzkes DR; AIDS Clinical Trials Group Study A5095 Team. Triple-nucleoside regimens versus efavirenz-containing regimens for the initial treatment of HIV-1 infection. N Engl J Med. 2004 Apr 29;350(18):1850-61. doi: 10.1056/NEJMoa031772. PMID 15115831
- [Result] Clifford DB, Evans S, Yang Y, Acosta EP, Goodkin K, Tashima K, Simpson D, Dorfman D, Ribaudo H, Gulick RM. Impact of efavirenz on neuropsychological performance and symptoms in HIV-infected individuals. Ann Intern Med. 2005 Nov 15;143(10):714-21. doi: 10.7326/0003-4819-143-10-200511150-00008. PMID 16287792
- [Result] Gulick RM, Ribaudo HJ, Shikuma CM, Lalama C, Schackman BR, Meyer WA 3rd, Acosta EP, Schouten J, Squires KE, Pilcher CD, Murphy RL, Koletar SL, Carlson M, Reichman RC, Bastow B, Klingman KL, Kuritzkes DR; AIDS Clinical Trials Group (ACTG) A5095 Study Team. Three- vs four-drug antiretroviral regimens for the initial treatment of HIV-1 infection: a randomized controlled trial. JAMA. 2006 Aug 16;296(7):769-81. doi: 10.1001/jama.296.7.769. PMID 16905783
- [Result] Ribaudo HJ, Kuritzkes DR, Schackman BR, Acosta EP, Shikuma CM, Gulick RM. Design issues in initial HIV-treatment trials: focus on ACTG A5095. Antivir Ther. 2006;11(6):751-60. PMID 17310819
- [Result] Kuritzkes DR, Ribaudo HJ, Squires KE, Koletar SL, Santana J, Riddler SA, Reichman R, Shikuma C, Meyer WA 3rd, Klingman KL, Gulick RM; ACTG A5166s Protocol Team. Plasma HIV-1 RNA dynamics in antiretroviral-naive subjects receiving either triple-nucleoside or efavirenz-containing regimens: ACTG A5166s. J Infect Dis. 2007 Apr 15;195(8):1169-76. doi: 10.1086/512619. Epub 2007 Mar 6. PMID 17357053
- [Result] Schackman BR, Ribaudo HJ, Krambrink A, Hughes V, Kuritzkes DR, Gulick RM. Racial differences in virologic failure associated with adherence and quality of life on efavirenz-containing regimens for initial HIV therapy: results of ACTG A5095. J Acquir Immune Defic Syndr. 2007 Dec 15;46(5):547-54. doi: 10.1097/qai.0b013e31815ac499. PMID 18193496
- [Result] Paredes R, Lalama CM, Ribaudo HJ, Schackman BR, Shikuma C, Giguel F, Meyer WA 3rd, Johnson VA, Fiscus SA, D'Aquila RT, Gulick RM, Kuritzkes DR; AIDS Clinical Trials Group (ACTG) A5095 Study Team. Pre-existing minority drug-resistant HIV-1 variants, adherence, and risk of antiretroviral treatment failure. J Infect Dis. 2010 Mar;201(5):662-71. doi: 10.1086/650543. PMID 20102271
- [Derived] Cardone KM, Dudek S, Keat K, Bradford Y, Cindi Z, Daar ES, Gulick R, Riddler SA, Lennox JL, Sinxadi P, Haas DW, Ritchie MD. Lymphocyte Count Derived Polygenic Score and Interindividual Variability in CD4 T-cell Recovery in Response to Antiretroviral Therapy. Pac Symp Biocomput. 2024;29:594-610. PMID 38160309
- [Derived] Li B, Veturi Y, Verma A, Bradford Y, Daar ES, Gulick RM, Riddler SA, Robbins GK, Lennox JL, Haas DW, Ritchie MD. Tissue specificity-aware TWAS (TSA-TWAS) framework identifies novel associations with metabolic, immunologic, and virologic traits in HIV-positive adults. PLoS Genet. 2021 Apr 26;17(4):e1009464. doi: 10.1371/journal.pgen.1009464. eCollection 2021 Apr. PMID 33901188
- [Derived] Leonard MA, Cindi Z, Bradford Y, Bourgi K, Koethe J, Turner M, Norwood J, Woodward B, Erdem H, Basham R, Baker P, Rebeiro PF, Sterling TR, Hulgan T, Daar ES, Gulick R, Riddler SA, Sinxadi P, Ritchie MD, Haas DW. Efavirenz Pharmacogenetics and Weight Gain Following Switch to Integrase Inhibitor-Containing Regimens. Clin Infect Dis. 2021 Oct 5;73(7):e2153-e2163. doi: 10.1093/cid/ciaa1219. PMID 32829410
- [Derived] Mollan KR, Smurzynski M, Eron JJ, Daar ES, Campbell TB, Sax PE, Gulick RM, Na L, O'Keefe L, Robertson KR, Tierney C. Association between efavirenz as initial therapy for HIV-1 infection and increased risk for suicidal ideation or attempted or completed suicide: an analysis of trial data. Ann Intern Med. 2014 Jul 1;161(1):1-10. doi: 10.7326/M14-0293. PMID 24979445
- [Derived] Lok JJ, Hunt PW, Collier AC, Benson CA, Witt MD, Luque AE, Deeks SG, Bosch RJ. The impact of age on the prognostic capacity of CD8+ T-cell activation during suppressive antiretroviral therapy. AIDS. 2013 Aug 24;27(13):2101-10. doi: 10.1097/QAD.0b013e32836191b1. PMID 24326304
- [Derived] Schouten JT, Krambrink A, Ribaudo HJ, Kmack A, Webb N, Shikuma C, Kuritzkes DR, Gulick RM. Substitution of nevirapine because of efavirenz toxicity in AIDS clinical trials group A5095. Clin Infect Dis. 2010 Mar 1;50(5):787-91. doi: 10.1086/650539. PMID 20121419